CLINICAL TRIAL: NCT06724133
Title: Relationship Among Oral Microbiome and NLRP3 Inflammatome and Colorectal Polyps
Status: Recruiting | Type: Observational
Sponsor: Limin Zhang (Other)
Responsible Party: Sponsor-Investigator, Limin Zhang, Dr, Shanghai 5th People's Hospital
Organization: Shanghai 5th People's Hospital (Other)
Other Study IDs: oral microbiome
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Search MeSH

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients diagnosed with colorectal polyps by enteroscopy in the gastroenterology department of our hospital were collected. For patients with two or more different types of histopathological examination results, all cases containing tubular adenoma, tubular villous adenoma and villous adenoma were classified into the adenoma group.
- Control group: Age - and sex-matched family members of the patient were selected, and no enteric-related diseases were detected by colonoscopy.

SUMMARY:
In this study, a case-control study was intended to establish a model for the combined diagnosis of colorectal polyps by detecting the expressions of oral and intestinal flora, ASC, Caspase-1, IL-1β and IL-18 in patients with colorectal polyps and healthy controls, as well as peripheral venous blood and intestinal tissue. To analyze the correlation between oral and intestinal specific flora and host inflammatory status, and explore the correlation between oral and intestinal flora, NLRP3 inflammatory complex, and colorectal polyps (pin-pin-two correlation), with a view to providing new biomarkers for the diagnosis and prognosis assessment of colorectal polyps from the perspective of oral and intestinal microorganisms and host immune inflammatory response. It also provides a new targeted treatment strategy for clinical prevention and treatment, and actively prevents the occurrence and development of colorectal polyp canceration.

ELIGIBILITY:
Inclusion Criteria:

* Case group: Patients diagnosed with colorectal polyps by enteroscopy in the gastroenterology department of our hospital were collected. For patients with two or more different types of histopathological examination results, all cases containing tubular adenoma, tubular villous adenoma and villous adenoma were classified into the adenoma group.

Control group: Age - and sex-matched family members of the patient were selected, and no enteric-related diseases were detected by colonoscopy.

Exclusion Criteria:

* a) The patient refuses to participate in the program; b) The patient has cognitive impairment and cannot cooperate with the researcher; c) Patients diagnosed with familial adenomatous polyposis or hereditary non-polyposis colorectal cancer, or with obvious familial genetic predisposition in the family, combined with other digestive system diseases and anorectal diseases; d) Infectious diseases; Such as respiratory tract, digestive tract, urinary system, reproductive system acute and chronic infection; e) Patients with a history of systemic disease: patients with serious lesions of heart, brain, liver, kidney and other important organs, such as organ dysfunction: cirrhosis, kidney failure, etc. (patients with severe heart, liver, and renal insufficiency); f) Immune diseases: such as connective tissue diseases, rheumatoid arthritis, etc.; g) Diseases of the blood system (have primary dyslipidemia, or have taken lipid-regulating drugs in the past 3 months); h) Patients with malignant tumors who have received radiotherapy and chemotherapy; i) a BMI of less than 18.5kg/m2 or a BMI of more than 32kg/m2 or severe malnutrition; j) Chronic metabolic diseases such as diabetes mellitus (including type 1 and type 2) and gout; k) Patients with a history of gastrointestinal surgery, or a history of intestinal surgery due to polyps or tumors; l) Pregnant and lactating women; m) Patients with edentulous jaws; n) Patients with a history of periodontal treatment in the past 6 months; o) Patients with fixed appliances in the mouth; p) Use probiotics, microbiotics, antibiotics, metformin, proton pump inhibitors, berberine and cathartic agents within the past 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with colorectal polyps and Healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Oral microbes | baseline
  Full-length 16S rRNA sequencing was used to investigate salivary samples.
fecal microbes | baseline
  Full-length 16S rRNA sequencing was used to investigate fecal samples.

SECONDARY OUTCOMES:
NLRP3 | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Fifth People's Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes